CLINICAL TRIAL: NCT06923644
Title: Targeted Precision Nutrition Strategy To Prevent Chronic Metabolic Diseases
Acronym: PRECINUT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Wageningen University and Research (Other); Health Holland (Other); TKI Agri & Food (Unknown); Nestle Health Science (Industry); Beneo GmbH (Industry); BARILLA G. e R. Fratelli S.p.A., Parma, Italy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NL87817.068.24
Record Dates: First submitted 2025-02-07; First posted 2025-04-11 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Obesity and Overweight; Pre-diabetic; Type 2 Diabetes Mellitus (T2DM)
Keywords: Dietary intervention trial; Precision nutrition; Tissue-specific insulin resistance; Body composition; Metabotyping; Glucose homeostasis; Cardiometabolic health; Insulin resistance; Metabolic phenotype
MeSH Terms: conditions — Obesity; Overweight; Glucose Intolerance; Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Precision Nutrition Group (PN) (Experimental): For a total duration of 12 months, participants in the Precision Nutrition (PN) Group will follow a diet tailored to their Metabotype, which is hypothesised to be optimal for them.
  Interventions: Other: Optimal Metabotype-specific diet
- Control Group (CN) (Experimental): For a total duration of 12 months, participants in the Control Group (CN) will be randomly assigned one of the diets optimised for a different Metabotype of the same sex, which is hypothesised to be suboptimal for them.
  Interventions: Other: Sub-optimal diet

INTERVENTIONS:
Other: Optimal Metabotype-specific diet — Following screening, baseline measurements, and determination of Metabotype, participants will be randomly assigned, using minimisation, to either the Precision Nutrition (PN) group or the Control (CN) group. The PN group will receive a diet hypothesised to be optimal for their specific Metabotype. All participants will adhere to their assigned diets for 12 months. Each Metabotype-specific diet will align with the Dutch Healthy Dietary Guidelines, while varying in macronutrient composition and quality.
  Arms: Precision Nutrition Group (PN)
Other: Sub-optimal diet — Participants randomised to the Control Group (CN), will be randomly assigned one of the two diets optimised for a different Metabotype of the same sex. The assigned CN Group diet will always have a macronutrient content and quality that is different than their hypothesised optimal diet. All diets will align with the Dutch Healthy Dietary Guidelines.
  Arms: Control Group (CN)

SUMMARY:
Nutrition is very important to keep blood sugar levels balanced. If blood sugar levels are too high, it can lead to diseases such as cardiovascular disease and type 2 diabetes (T2DM). Therefore, adjusting what one eats, also called a diet or nutritional intervention, can help prevent these diseases. However, not everyone responds the same to a diet. In about 30% of people, a diet does not work as hoped. This can be due to various reasons, such as a person's metabolism, genetic predisposition, the composition of the food one eats, or the bacteria in the intestines. Everyday things like sleep, stress, and movement also play a role. The investigators used a computer model to classify people with overweight and obesity into groups based on these factors. The investigators call such a group a 'Metabolic Phenotype', or in short 'Metabotype'. Based on the Metabotype, a personalised diet was developed (personalised nutrition intervention) that may better suit each person's unique situation.

The investigators hypothesize that a precision nutrition intervention, tailored to Metabotypes identified through unsupervised clustering (using the aforementioned computer model) of predefined, accurate features related to cardiometabolic health-specifically, tissue-specific glucose and lipid metabolism and detailed body composition-will enhance blood glucose homeostasis, reduce cardiometabolic risk, and improve adherence to the intervention and mental well-being, compared to population-based dietary guidelines. The present project will contribute to targeted and efficient precision-based dietary strategies for individuals at increased risk of T2DM.

DETAILED DESCRIPTION:
Objective:

Our study aims to identify unique Metabotypes among individuals with overweight and obesity and assess their response to a 1-year precision dietary macronutrient modulation. The objective is to provide proof-of-concept that this approach improves glucose homeostasis, dietary adherence, and psychosocial well-being compared to population-based dietary guidelines.

Study design:

Two-centre dietary intervention study with a double-blind, randomised controlled parallel design, based on participants' Metabotype and hypothesized optimal diet. Participants' Metabotype and intervention arm will be blinded to the participants and researchers. Metabotypes were identified through hierarchical clustering of Principal Components (HCPC) using baseline data from The Maastricht Study (participant demographics, body composition, glucose- and insulin metabolism), whereafter clusters were cross-validated in independent cohorts. Based on a combination of post-hoc analyses of dietary intervention trials and literature, the optimal dietary macronutrient composition was determined for these Metabotypes.

Study population:

In total 240 men and women with overweight and obesity (age 40-75 years, BMI 25-40 kg/m2) will be included. Further details on in- and exclusion criteria will be described under ''Eligibility''. Following screening and baseline measurements, for each eligible participant, a classification algorithm will determine the participants' Metabotype cluster (one of three possible Metabotypes for each sex).

Intervention:

Following screening, baseline measurements, and determination of Metabotype, participants will be randomly assigned, using minimization, to either the Precision Nutrition (PN) group or the Control (CN) group. The PN group will receive a hypothesized optimal diet for their specific Metabotype, while the control group will be randomly assigned one of the diets optimized for a different Metabotype of the same sex. All participants will follow their assigned diets for 12 months, with each diet conforming to the Dutch healthy dietary guidelines. Participants will receive regular dietary consultation, and meal plans including variation lists to guide them with their dietary intake during the intervention.

Main study parameters/endpoints:

Extensive characterization will be done before, during, and after the intervention. Primary outcome measure is whole-body insulin sensitivity (Matsuda index) assessed by means of a 7-point oral glucose tolerance test (OGTT). Secondary outcomes include glycaemic variability, mean glucose levels, fasting lipid profiles, body composition, blood pressure, gene and protein expression of adipose tissue, microbial composition and functionality, metabolomics, physical activity, adherence to dietary recommendations, (mental) well-being, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with a BMI ≥25 to <40 kg/m2
* Classification possible to one of the investigational metabolic phenotypes according to the classification algorithm.
* Weight stability for at least 3 months (+/- 3 kg)

Exclusion Criteria:

Diseases

* (Pre-)diagnosis of type 1 or type 2 diabetes mellitus (i.e., FPG ≥ 7,0 mmol/L) and HbA1c ≥ 6,5% (48 mmol/mol)
* Renal or hepatic malfunctioning (pre-diagnosis or determined based on ALAT and creatinine values)
* Gastrointestinal diseases or abdominal surgery (allowed i.e.:

appendectomy, cholecystectomy)

* Food allergies, intolerances (including gluten/lactose intolerance) and/or eating disorders interfering with the study
* Cardiovascular diseases (e.g., heart failure) or cancer (e.g., noninvasive skin cancer allowed)
* High systolic blood pressure (untreated >160/100 mmHg, drug-regulated >140/90 mmHg)
* Diseases affecting glucose and/or lipid metabolism (e.g., pheochromocytoma, Cushing's syndrome, acromegaly)
* Diseases with a life expectation shorter than 5 years
* Major mental disorders
* Drug treated thyroid diseases (well substituted hypothyroidism is allowed inclusion)
* Other physical/mental conditions that may interfere with study outcomes

Medication

* Medication known to interfere with study outcomes (e.g., PPAR-α or PPAR-γ agonists (fibrates), sulfonylureas, biguanides, α-glucosidaseinhibitors, thiazolidinediones, repaglinide, nateglinide, insulin, and chronic use of NSAIDs)
* Use of certain anticoagulants other than acetylsalicylic acid
* Use of antidepressants (stable use ≥ 3 months prior to and during study allowed)
* Use of statins (stable use ≥ 3 months prior to and during study allowed)
* Chronic corticosteroids treatment (>7 consecutive days of treatment)
* Use of antibiotics within 3 months prior to the study

Lifestyle

* Participation in regular sports activities (moderate-to-vigorous physical exercise >4 hours per week)
* Having a restricted dietary pattern interfering with the study diets (e.g., vegetarian, vegan, Atkins diet and/or other special diets)
* Plans to lose or gain more than 5% body weight
* Abuse of alcohol (alcohol consumption >14 units/week) and/or drugs (cannabis included)
* Not willing to limit alcohol consumption to 7 drinks per week
* Regular smoking (including use of e-cigarettes and vapes)
* Use of strong vitamins or other dietary supplements (e.g., pre- or probiotics) expected to interfere with the study outcomes

Other

* Metabotype classification is not possible
* Pregnant or lactating women, or women who are planning to become pregnant
* Inability to comply with the study diet
* Blood donation within the last 3 months
* Participation in possibly interfering studies within the last 3 months
* Inability to understand study information and/or communicate with staff
* Unwillingness to be randomised or sign informed consent
* Unwillingness to save data for 15 years
* Deemed unsuitable for participation in the trial, for any reason, as judged by the research physician or principal investigator

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 240 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Matsuda Index | Change from baseline at month 6 and month 12 following dietary intervention.
  The primary objective of this study is to evaluate the effect of a 12-month Metabotype-targeted diet (PN) versus a non-targeted diet (CN) on whole-body insulin sensitivity (Matsuda Index; marker of whole-body fasting and postprandial insulin sensitivity). This will include within group post-hoc testing. The primary outcome measure will be assessed by means of a 7-point oral glucose tolerance test (OGTT), and calculated as follows: [10,000 / square root of [fasting plasma glucose (mg/dL) × fasting insulin (mU/L)] × [mean glucose (mg/dL) x mean insulin (mU/L)]].

SECONDARY OUTCOMES:
Glucose tolerance | Change from baseline at month 6 and month 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. Determined by 2-hour plasma glucose values (mmol/L) during an oral glucose tolerance test (OGTT).
Disposition Index (DI) | Change from baseline at month 6 and month 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. The Disposition Index is a composite marker of first phase insulin secretion and insulin sensitivity during a 2-hour 7-point oral glucose tolerance test (OGTT). Disposition index will be calculated as follows: [Insulin sensitivity index (ISI) * (AUC30 min insulin / AUC30 min glucose)], where AUC30 min is the area under the curve between 0 and 30 minutes of the OGTT for insulin (pmol/l) and glucose (mmol/l), respectively, and ISI is defined as: [10,000 ÷ square root of (fasting plasma glucose (mmol/l) x fasting insulin (pmol/l)) x (mean glucose (mmol/l) x mean insulin (pmol/l))]. Higher values represent a higher insulin sensitivity.
HOMA-IR | Change from baseline at month 6 and month 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. HOMA-IR is a fasting measure for insulin resistance, which can be calculated as follows: HOMA-IR = (Fasting plasma glucose (mmol/L) * Fasting Insulin (mU/L)) / 22.5. Higher values represent a higher degree of insulin resistance. Determined in plasma during a 2-hour, 7-points oral glucose tolerance test (OGTT).
Muscle insulin sensitivity (MISI) | Change from baseline at month 6 and month 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. Determined during a 2-hour, 7-point oral glucose tolerance test (OGTT). The muscle insulin sensitivity index (MISI) will be calculated as follows: MISI (mmol/l/min/pmol/l) = (dG/dt) / mean plasma insulin concentration (pmol/l) during OGTT. Here, dG/dt is the rate of decay of plasma glucose concentration (mmol/L) during the OGTT, calculated as the slope of the least square fit to the decline in plasma glucose concentration from peak to nadir. Higher values represent higher muscle insulin sensitivity.
Hepatic insulin resistance (HIRI) | Change from baseline at month 6 and month 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. Determined during a 2-hour, 7-point oral glucose tolerance test (OGTT). The hepatic insulin resistance index (HIRI) will be calculated using the square root of the product of the area under curves (AUCs) for plasma glucose and insulin during the first 30 min of the OGTT - i.e., square root (glucose0-30 [AUC in mmol/l·h] · insulin 0-30 [AUC in pmol/l·h). Higher HIRI values represent lower hepatic insulin sensitivity.
Adipose tissue insulin sensitivity (ATIRI) | Change from baseline at month 6 and month 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. The Adipose Tissue Insulin Resistance Index (ATIRI) is an indicator of the degree of insulin resistance in adipose tissue. Determined during a 2-hour, 7-point oral glucose tolerance test (OGTT), using fasting plasma insulin and free fatty acids (FFA) concentrations. ATIRI is calculated as: fasting FFA (mmol/L) * fasting Insulin (pmol/L. Higher ATIRI values represent lower adipose tissue insulin sensitivity.
Insulinogenic Index (IGI) | Change from baseline at month 6 and month 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. Determined during a 2-hour, 7-point oral glucose tolerance test (OGTT). The Insulinogenic Index (IGI) is a measure used to assess the early insulin response of the pancreas to a glucose load. IGI is calculated as: Plasma Insulin 0 - 30 [AUC in pmol/L x min] / Glucose 0 - 30 [AUC in mmol/L x min]. Higher IGI values represent a higher proportional secretion of insulin in response to insulin, indicative of a proportional increased pancreatic secretion of insulin.
HOMA-β | Change from baseline at month 6 and month 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. Determined during a 2-hour, 7-point oral glucose tolerance test (OGTT), based on fasting plasma glucose and fasting insulin levels. Homeostatic Model Assessment of Beta-cell function (HOMA-β) is a mathematical model used to estimate the function of pancreatic beta-cells, which are responsible for producing insulin. HOMA-β is calculated as: 20 × (fasting insulin (mU/L) / (fasting glucose (mmol/L) - 3.5). Normal values are ~100, higher values are indicative of increased Beta-cell activity, while lower values are indicative of decreased Beta-cell activity.
Circulating hormones such as Insulin | Change from baseline at month 6 and month 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. Circulating hormones such as insulin are determined in plasma during a 2-hour, 7-point oral glucose tolerance test (OGTT).
Body composition | Change from baseline at month 6 and month 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. Body composition such as the Android/Gynoid fat mass ratio (unitless) will be determined by using a dual-energy X-ray absorptiometry scan (DXA).
Waist circumference | Change from baseline at month 6 and month 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. Waist circumference in centimeters.
Hip circumference | Change from baseline at month 6 and month 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. Hip circumference in centimeters.
Waist-to-hip ratio (WHR) | Change from baseline at month 6 and month 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. Waist circumference in centimeters, divided by the hip circumference in centimeters, expressed as a unitless ratio.
Subcutaneous adipose tissue gene expression | Change from baseline at month 6 and month 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. Subcutaneous adipose tissue biopsies will be taken for gene expression analysis. Biopsies will only be obtained in a sub-group of participants at the MUMC+, none will be obtained from participants at WUR.
Subcutaneous adipose tissue protein expression | Change from baseline at month 6 and month 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. Subcutaneous adipose tissue biopsies will be taken for protein expression analysis. Biopsies will only be obtained in a sub-group of participants at the MUMC+, none will be obtained from participants at WUR.
Blood pressure | Change from baseline at month 6 and month 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. Systolic and diastolic blood pressure in mmHg.
Mean 24h glucose concentrations | Change from baseline at month 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. For a 14-day period at the beginning and end of the intervention, mean 24-hour glucose levels will be monitored in all participants with a glucose sensor (FreeStyle libre 2, Research CGM, Abbot).
Glucose incremental area under the curve (iAUC) | Change from baseline at month 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. For a 14-day period at the beginning and end of the intervention, 24-hour glucose levels will be monitored in all participants with a glucose sensor (FreeStyle libre 2, Research CGM, Abbot). The net incremental area under the curve (iAUC) will be calculated by the trapezoid rule, using fasting glucose value as baseline. The iAUC provides a summary measure of the net increase in glucose levels above the fasting level during the 24-hour period.
The frequency of hypo- and hyperglycemia | Change from baseline at month 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. For a 14-day period at the beginning and end of the intervention, 24-hour glucose levels will be monitored in all participants with a glucose sensor (FreeStyle libre 2, Research CGM, Abbot). The frequency of hypo- and hyperglycaemia will be monitored and defined as occurrences of a glucose level of ≥10.0 mmol/l for hyperglycaemia, whilst hypoglycaemia will be defined as a glucose concentration ≤ 3.9 mmol/l.
Mean Amplitude of Glucose Excursions (MAGE) | Change from baseline at month 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. For a 14-day period at the beginning and end of the intervention, 24-hour glucose levels will be monitored in all participants with a glucose sensor (FreeStyle Libre 2, Research CGM, Abbott).
  The Mean Amplitude of Glucose Excursions (MAGE) will be calculated as the average of significant glucose fluctuations (excursions) above or below the mean glucose level. MAGE quantifies glycemic variability and is expressed in mmol/L.
Time in Range (TIR) | Change from baseline at month 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. For a 14-day period at the beginning and end of the intervention, 24-hour glucose levels will be monitored in all participants with a glucose sensor (FreeStyle Libre 2, Research CGM, Abbott).
  The Time in Range (TIR) will be defined as the percentage of time spent within the target glucose range of 3.9-10.0 mmol/L. Time spent below 3.9 mmol/L (time below range, TBR) and above 10.0 mmol/L (time above range, TAR) will also be calculated as secondary metrics.
Coefficient of Variation (CV%) | Change from baseline at month 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. For a 14-day period at the beginning and end of the intervention, 24-hour glucose levels will be monitored in all participants with a glucose sensor (FreeStyle Libre 2, Research CGM, Abbott).
  The Coefficient of Variation (CV%) will be calculated as the standard deviation of glucose divided by the mean glucose level, multiplied by 100. CV% expresses glucose variability as a percentage and reflects overall glycemic stability, with a CV% > 36% considered indicative of high variability.
Standard Deviation (SD) of Glucose Levels | Time Frame: Change from baseline at month 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. For a 14-day period at the beginning and end of the intervention, 24-hour glucose levels will be monitored in all participants with a glucose sensor (FreeStyle Libre 2, Research CGM, Abbott).
  The Standard Deviation (SD) of glucose levels will be calculated as a measure of glycemic variability around the mean glucose concentration. A higher SD indicates greater glucose fluctuation and variability throughout the monitoring period.
The duration of hypo- and hyperglycemia | Change from baseline at month 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. For a 14-day period at the beginning and end of the intervention, 24-hour glucose levels will be monitored in all participants with a glucose sensor (FreeStyle libre 2, Research CGM, Abbot). The duration of hypo- and hyperglycaemia will be monitored and defined as time spent with a glucose level of ≥10.0 mmol/l for hyperglycaemia, whilst hypoglycaemia will be defined as a glucose concentration ≤ 3.9 mmol/l.
Gut microbial composition | Change from baseline at month 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. Faecal samples to be used for analysing microbiota composition will be collected.
Circulating SCFA | Change from baseline at month 6 and month 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. Circulating Short Chain Fatty Acids (SCFAs) are determined in plasma during a 2-hour, 7-point oral glucose tolerance test (OGTT).
Targeted plasma metabolomics | Baseline
  At baseline, a fasting blood sample will be collected during the oral glucose tolerance test (OGTT) for determination of the Metabotypes' metabolomics profile (Nightingale).
Circulating lipids such as FFA | Change from baseline at month 6 and month 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. Circulating lipids such as Free Fatty Acids (FFA) are determined in serum during a 2-hour, 7-point oral glucose tolerance test (OGTT).
Circulating inflammatory markers such as CRP | Change from baseline at month 6 and month 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. Circulating inflammatory markers such as C-Reactive Protein (CRP) are determined in plasma during a 2-hour, 7-point oral glucose tolerance test (OGTT).
Circulating HbA1c | Change from baseline at month 6 and month 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. Circulating Hemoglobin A1c (HbA1c) is determined in plasma during a 2-hour, 7-point oral glucose tolerance test (OGTT).
Physical activity | Change from baseline at month 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. Physical activity patterns will be monitored continuously with the ActivPAL device during a 14-day period at baseline and at the end of the intervention.
Self-reported self-efficacy | Change from baseline at month 6 and 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. Self-efficacy with regard to health behaviour is measured by the 13-item PAM-13 (Patient Activation Measurement questionnaire). Score ranges from 0-100, higher scores indicate a greater self-efficacy.
Self-reported context-sensitive positive health | Change from baseline at month 1 and 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. Positive health is measured by the 23-item Context-sensitive Positive Health Questionnaire (CPHQ), which is a newly developed questionnaire still in the validation phase. Score ranges from 0-100, higher scores indicate a greater positive health.
Self-reported mood | Change from baseline at month 6 and 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. Potential positive impacts on mood by the intervention are measured by the 20-item PANAS, resulting in a positive mood score (10-50; higher scores representing higher levels of positive mood), and negative mood score (10-50; lower scores representing lower levels of negative mood).
Self-reported stool consistency | Change from baseline at month 1 and 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. Stool consistency is measured by the Bristol Stool Chart (BSC). Score ranges from 1-7, wherein 1-2 indicates constipation, 3-4 normal stool, and 5-7 diarrhoea.
Self-reported fatigue | Change from baseline at month 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. Physical and mental fatigue are assessed using the 14-item Chalder fatigue scale. Scores range 0-42, wherein higher scores indicate increasing fatigue severity.
Self-reported health-related quality of life | Change from baseline at month 1 and 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. Health-related quality of life is measured by the 6-item EQ5-D is a short scoring tool for mobility, self-care, daily activities, pain/discomfort and fear/depression, complementary to the CPHQ. The score consists of a health index (ranging from -0.59 to 1.00, with 1 being perfect health) based on aforementioned five dimensions and a visual analog scale (VAS) from 0 to 100 to assess self-rated health.
Self-reported positive health | Change from baseline at month 1 and 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. Positive health is measured by the 17-item IPH-17, which is a shortened positive health questionnaire, complementary to the CPHQ. Scores range from 17-85, higher scores indicate more concerns about own health.
Adherence to dietary recommendations | 12-months, continuously throughout the study
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. During the 12-month intervention period, dietary compliance will be assessed before each planned visit at 1, 3, 6, 9 and 12 months. In short, roughly two weeks before each visit, participants will receive a prompt to record their food intake on two week-days and one weekend-day via Traqq App. These recording days will be automised, unannounced and non-consecutive.
Self-reported mental health | Change from baseline at month 6 and 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. Mental wellbeing is assessed using the RAND-36. Scored from 0 to 100, higher scores represent better mental health.
Self-reported perceived stress | Change from baseline at month 6 and 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. Perceived stress is measured with the 10-item Perceived Stress Scale (PSS10). Scores range from 0-40, higher scores represent higher levels of perceived stress.
Self-reported gastrointestinal health | Change from baseline at month 1 and 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. Gastrointestinal symptoms are assessed by the 15-item Gastrointestinal Symptom Rating Scale (GSRS). Scores range from 15-105, wherein higher scores indicate more severe discomfort.
Self-reported sleep quality | Change from baseline at month 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. Sleep quality is assessed with the 10-item Pittsburgh Sleep Quality Index. Scores range 0-21, higher scores indicate worse sleep quality.
Self-reported daytime sleepiness | Change from baseline at month 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. Daytime sleepiness is assessed with the 8- item Epworth Sleepiness scale. Scores range 0-24, higher scores indicate greater daytime sleepiness.
Self-reported chronotype | Change from baseline at month 12 following dietary intervention.
  Optimal (PN) versus sub-optimal (CN) diet, including within group post-hoc testing. The Munich Chronotype Questionnaire (MCTQ) assesses an individual's chronotype (biological sleep-wake preference) based on actual sleep behaviour on workdays and free days. MCTQ determines chronotype based on the midpoint of sleep on free days (MSF; hh:mm, 24-hour format)), adjusted for sleep debt (MSFsc; hh:mm, 24-hour format), and social jetlag (SJL; hh:mm, 24-hour format), where later MSFsc indicates an evening type and higher SJL reflects circadian misalignment.
DNA analysis | Baseline
  Buffy coats will be collected for DNA analysis, pre-intervention only, exploratory objective.

OTHER OUTCOMES:
Baseline characteristics | Baseline
  Baseline characteristics (age, sex, ethnicity, lifestyle, socioeconomic status, medical history, medication use, family composition and history of T2DM, and menopausal state) will also be recorded, for the purpose of screening, metabolic classification and potential post-hoc analysis.
Metabotype cluster | Baseline, and change from baseline at month 6 and month 12 following dietary intervention.
  The Metabotype cluster (one of three possible groups for each sex) will be assessed at three time points. Namely, baseline, at 6 months and at 12 months. To determine the Metabotype, several outcome measures derived from the OGTT and anthropometrics will be aggregated by the described classification algorithm (see study description).
Capillary Blood Samples (CBS) | Baseline and following 12 month dietary intervention.
  Capillary Blood Samples (CBS) samples will be obtained via fingerpick parallel to the venous fasting blood sample collected during the oral glucose tolerance test (OGTT). These samples will be analyzed to explore the feasibility of developing a simplified classification algorithm for determining Metabotype, providing a potentially more accessible and less invasive diagnostic approach. CBS will only be obtained in a sub-group of participants at the MUMC+, none will be obtained from participants at WUR.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen E Blaak, Prof. Dr. Ir., Principal Investigator — Maastricht University Medical Center
Locations (2):
- Netherlands (2):
  - Maastricht University Medical Center, Department of Human Biology, NUTRIM Institute of Nutrition and Translational Research in Metabolism, Maastricht
  - Wageningen University and Research, Division of Human Nutrition, Wageningen

IPD SHARING:
Plan to Share IPD: Yes
Once the corresponding article is published and/or the project is finished, (part of) our metadata will be accessible for further research and verification. Interested researchers can submit a data request by means of a synopsis, this is necessary to prevent inappropriate use of data. A designated committee consisting of the project leader and the steering committee will decide on the approval of future requests (synopsis) for data access. At a minimum, the synopsis must show that the applicant's intended purpose and method of operation comply with the PRECINUT Data Terms of Use (see also access criteria), which have yet to be determined by the steering committee.
  Study participants will be provided with a participant number, which can only be connected to personal data via the informed consent form. The informed consent forms are only stored at the respective research sites separately (MUMC+/WUR), and will not be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Possibly, based on guidelines in the consortium agreement, the steering committee could agree on an embargo period, which could delay the accessibility of (part of) the data. One of the reasons for delayed data access may be the application for IP rights and marketing of the acquired knowledge (by consortium partners).
Access Criteria: * The purpose of data access is limited to scientific purposes and may not be used for commercial purposes;
  * The purpose of the data request must be of public interest. Research questions of the data access applicant must be related to the research topic of the original study;
  * The dataset must not be linked to an external dataset (for privacy reasons);
  * Use of the dataset is not infinite, but only for a predetermined period, a time interval required for analyses of data up to a maximum of 3 months (and once for this specific question by this applicant);
  * A small fee is requested for (re)use of the data. This fee will cover the additional costs associated with assessing the request and distributing the data;
  * If the purpose of data access is scientific publication, agreements must be made in advance on co-authorship, access to the final manuscript and the possibility of stopping the publication of data up to a period of 3 months if no agreement can be reached between parties.